CLINICAL TRIAL: NCT04710264
Title: An Observational Cohort Study to Evaluate the Expression Profiles of Oocyte-potency-related Genes in Ovarian Cumulus Cells From Patients Treated by Intracytoplasmic Sperm Injection (ICSI) That Are Treated With Recombinant Gonadotropins
Brief Title: Aurora Test for Patients Treated With Recombinant Gonadotropins
Acronym: AURORA-REC
Status: Completed | Type: Observational
Sponsor: Fertiga, Belgium (Industry)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020.Aurora-Rec
Record Dates: First submitted 2021-01-09; First posted 2021-01-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- recombinant hFSH: Patient stimulated with recombinant hFSH
  Interventions: Other: AURORA-Rec
- recombinant hFSH : r-hLH: Patient stimulated with recombinant hFSH : r-hLH ratio 2:1
  Interventions: Other: AURORA-Rec

INTERVENTIONS:
Other: AURORA-Rec — Explorative study of cumulus cells gene expression in relation to the patient treatment and oocyte competence.

SUMMARY:
This is an observational study. The main aim is to determine the expression of potential biomarker genes in the cumulus cells isolated from individual oocytes in two patient cohorts: recombinant human Follicle Stimulating Hormone(hFSH) and recombinant hFSH:human Luteinizing Hormone(r-hLH) ratio 2:1. Algorithms from gene combinations will be identified that predict embryo quality and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients are between 22-38 years old
* BMI between 17-33
* provide written informed consent
* Patients undergoing a first or second ICSI treatment cycle.
* Patients will be treated by ICSI (intracytoplasmic sperm injection)
* Patients agree that the oocytes will be denuded for cumulus testing and agree to the single blastocyst transfer.
* Patients must be predicted good ovarian responders (AMH 1-4,7 ng/ml) with 7-18 follicles of minimum 10-11 mm on trigger day (oocyte retrieval minus 2 days (OR -2)) by ultrasound following ovarian stimulation with r-hFSH or r-hFSH with r-hLH in a Gonadotropin-releasing hormone (GnRH) antagonist protocol (starting dose recombinant Follicle Stimulating Hormone (rFSH) between 150-225 IU)
* HCG trigger after stimulation (r-hCG)

Exclusion Criteria:

* Women with less than 7 or more than 18 follicles at Day -2 or -3 measured by ultrasound
* Women with history of poor oocyte maturation or known maturation defect
* Irregular menstrual cycle (< 24 or > 35 days)
* BMI < 17 or > 33
* Smoking > 10 cigarettes per day.
* Known low ovarian response based on Bologna criteria
* Combined use of urinary and recombinant gonadotropins in the current cycle
* Patients with severe endometriosis ≥ III (AFS classification)
* Polycystic ovary syndrome (PCOS), defined by revised criteria American Society for Reproductive Medicine (ASRM) European Society of Human Reproduction and Embryology (ESHRE) 2018
* Patient included in any other study
* Patient scheduled for preimplantation genetic testing (PGT)
* Testicular sperm extraction (TESE) or extreme oligo-astheno-teratozoospermia (OAT) with sperm count below 100.000/ml.

Ages: 22 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients for this study must be between 22-38 years of age, have a good ovarian reserve and response, and need to be naïve to IVF/ ICSI or have only one prior ICSI cycle. Only patients with 7-18 follicles at the end of ovarian stimulation will be allowed to enter the study on the day of decision of hCG injection (or the day before). Patients with fewer than 7 oocytes will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Normalized messenger ribonucleic acid (mRNA) expression | 3 years after study start
  Normalized mRNA levels of biomarker genes that are assessed in cumulus cells by reverse transcription quantitative Polymerase Chain Reaction (RT-qPCR) for each oocyte.

SECONDARY OUTCOMES:
Meiosis II Oocyte rate | Day 0 of embryo collection
  The number of meiosis II oocytes (nominator) divided by the total number of oocytes retrieved (denominator)
Normal fertilization rate | Day 1 of embryo culture
  The number of fertilized oocytes on Day 1 (presence of 2 pronuclei (2PN) and the second polar body (2PB) assessed at 17 ± 1 h postinsemination, as a function of all cumulus-oocytes complexes (COCs) inseminated
Day 5 good-quality embryo rate | Day 5 of embryo culture
  Defined as the proportion of 2PN zygotes which are good-quality blastocysts on Day 5
Embryo utilization rate | Day 5 of embryo culture
  Defined as the number of embryos (or blastocysts) suitable for transfer or cryopreservation as a function of the number of normally fertilized (2PN) oocytes observed on Day 1
Biochemical pregnancy rate | Day 10 after embryo transfer
  A pregnancy diagnosed only by the detection of beta human chorionic gonadotropin (hCG) in serum or urine
Fetal heart beat positive implantation rate | Week 5-6 after embryo transfer
  Rate refers to the proportion of fetal heartbeats detected relative to the number of embryos transferred
Clinical pregnancy rate | Week 5-6 after embryo transfer
  Pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat in gestational week 6 to 8
Ongoing pregnancy rate | Week 10-11 after embryo transfer
  The presence of gestational sacs with fetal heart beat detected by transvaginal ultrasound examination in gestational week 10 to 11
Miscarriage rate | Week 12 after embryo transfer
  The spontaneous loss of an intra-uterine pregnancy prior to 22 completed weeks of gestational age. In this study we capture spontaneous miscarriage till gestational week 12.

OTHER OUTCOMES:
Cumulative ongoing pregnancy rate | 3 years after study start
  The accumulated ongoing pregnancy after fresh and frozen-warmed embryo transfers within one stimulation cycle. Pregnancy with detectable heart rate at ≥ 12 weeks gestation after the completion of the first transfer
Live Birth rate | Week 24-42 after embryo transfer
  is defined as the birth of at least one newborn after 24 weeks gestation that exhibits any sign of live (twins will be a single count)
Cumulative Live Birth rate | 3 years after study start
  The number of deliveries with at least one live birth resulting from one initiated or aspirated artificial reproductive technologies (ART) cycle, including all cycles in which fresh and/or frozen embryos are transferred, until one delivery with a live birth occurs or until all embryos are used, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adriaenssens T, Van Vaerenbergh I, Van Leuven W, Coucke W, Montenegro S, Zheng W, D'Hooghe T, Van Landuyt L, De Munck N, Van Hecke E, Smitz J, Rosenthal A, Blockeel C. Live birth in patients stimulated with r-hFSH or r-hFSH: r-hLH is strongly associated with cumulus cell derived gene expression models. Reprod Biol Endocrinol. 2025 Nov 22;23(1):163. doi: 10.1186/s12958-025-01480-2. PMID 41275247